CLINICAL TRIAL: NCT02014051
Title: Phase I Clinical Trial of SyB C-1101 in Patients With Myelodysplastic Syndrome
Brief Title: Safety and Pharmacokinetics Study of SyB C-1101 in Patients With Recurrent/Relapsed or Refractory Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012002
Record Dates: First submitted 2013-12-01; First posted 2013-12-17 (Estimated); Results first posted 2016-09-14 (Estimated); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes

ARMS (1):
- SyB C-1101 (Experimental)
  Interventions: Drug: SyB C-1101

INTERVENTIONS:
Drug: SyB C-1101 — SyB C-1101（rigosertib sodium） will be administered to two cohorts at either 280 mg/day or 560 mg/day.
  The dose will be administered orally twice daily for 14 consecutive days, followed by 7-day observation period. The treatment period of 21 days (14 days of administration + 7 days of observation) constitutes 1 cycle.
  The study will involve treatment through the second cycle, but treatment can be continued for 3 or more cycles if conditions for continued administration are satisfied. However, treatment will be limited to a maximum of 6 cycles including the first cycle.

SUMMARY:
The purpose of this study is to investigate tolerability when SyB C-1101 is orally administered twice daily for 14 consecutive days to the patients with recurrent/relapsed or refractory myelodysplastic syndrome, to determine the dose-limiting toxicity and maximum tolerated dose, and to estimate the recommended dose for phase II studies. Pharmacokinetics and antitumor effects will also be investigated.

DETAILED DESCRIPTION:
In Cohort 1, SyB C-1101 280 mg/dose group, Participants will be administered 280 mg/dose of SyB C-1101 twice daily orally for 14 consecutive days, followed by 7-day observation period.

In Cohort 2, SyB C-1101 560 mg/dose group, Participants will be administered 560 mg/dose of SyB C-1101 twice daily orally for 14 consecutive days, followed by 7-day observation period.

In both Cohorts, the treatment period of 21 days constitutes 1 cycle, and the treatment was allowed for up to cycles. The participants received SyB C-1101 only once daily on Day 1 and Day 14 of Cycle 1 for the investigation of the pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy the following conditions listed below:

1. Patients who have been histologically documented or cytologically confirmed with myelodysplastic syndrome (MDS), and who have been found to meet any of the following criteria on the basis of the World Health Organization (WHO) classification or the French-American-British (FAB) classification.

   * Refractory Anemia (RA)* (< 5% myeloblasts, < 15% ringed sideroblasts)
   * RA with Ring Sideroblasts (RARS)* (< 5% myeloblasts, >= 15% ringed sideroblasts)
   * RA with Excess of Blasts-1(RAEB-1)(5% to 9% myeloblasts)
   * RAEB-2 (10% to 19% myeloblasts)
   * RAEB-t (20% to 29% myeloblasts or < 25,000/mm^3 peripheral leukocytes)
   * Chronic myelomonocytic leukemia (CMML) (10% to 19% myeloblasts, >= 1,000/mm^3 peripheral monocytes, < 13,000/mm^3 leukocytes) * RA and RARS patients should have 2 or more units of erythrocyte transfusion within 8 weeks.
2. Patients with a low value in at least one blood cell lineage (having at least one of the following cytopenias).

   * Neutrophils : < 1,800/mm^3
   * Platelets : < 100,000/mm^3
   * Hemoglobin : < 10 g/dL
3. Patients with a previous history of chemotherapy (including immunosuppressive therapy, anabolic steroid and lenalidomide) for the target disease who meet any of the following criteria.

   * Patients who have not achieved complete remission, partial remission, or hematologic improvement.*
   * Patients with recurrence/relapse after complete remission, partial remission, or hematologic improvement.*
   * Patients with intolerability that has led to discontinuation of treatment because of the development of liver dysfunction, kidney dysfunction, etc., after the start of treatment. *Proximate therapeutic efficacy judged under International Working Group (IWG) 2006 criteria.
4. For the patients who have received chemotherapy such as immunosuppressive therapy, anabolic steroid and lenalidomide, the patients should have not been treated for four weeks or longer after the end of the previous therapy and be judged to have no residual effects (antitumor effects) from the previous therapy.
5. Patients who can be expected to survive at least three months or longer.
6. Patients at least 20 years old (when informed consent is obtained).
7. Patients who have score of 0 to 2 in The Eastern Cooperative Oncology Group (ECOG) Performance Status (PS).
8. Patients with adequate function in major organs (heart, lungs, liver, kidneys, etc.).

   * Aspartate aminotransferase (AST) : no greater than 3.0 times the upper boundary of the reference range at each institution
   * Alanine aminotransferase (ALT) : no greater than 3.0 times the upper boundary of the reference range at each institution
   * Total bilirubin: no more than 1.5 times the upper boundary of the reference range at each institution
   * Serum creatinine: no more than 1.5 times the upper boundary of the reference range at each institution
   * ECG: no abnormal findings requiring treatment
   * Echocardiography: no abnormal findings requiring treatment
9. Patients who personally signed an informed consent document for participation in this study.

Exclusion Criteria:

Patients who satisfy any of the following conditions will not be enrolled in the study.

1. Patients with anemia caused by factors other than MDS (hemolytic anemia, gastrointestinal (GI) bleeding, etc.)
2. Patients with hypoplasia MDS (< 10% osteocyte density)
3. Patients who have undergone treatment for an active malignant tumor within the past year (except basal cell or squamous cell skin cancer, or primary squamous cell carcinoma of the cervix or noninvasive breast cancer).
4. Patients who have been administered a cytokine preparation such as G-CSF (granulocyte-colony stimulating factor), erythropoietin, etc. within 14 days of tests for enrollment of the study.
5. Patients with obvious infectious diseases (including viral infections).
6. Patients with serious complications (liver failure, renal failure, etc.).
7. Patients with a complication or previous history of serious heart disease (myocardial infarction, ischemic heart disease, etc.) within the past two years before enrollment, and with cardiac arrhythmia requiring treatment.
8. Patients with a serious gastrointestinal condition (severe or significant nausea/vomiting, diarrhea, etc.)
9. Patients who are positive for the Hepatitis B surface (HBs) antigen or HIV antibodies.
10. Patients with serious bleeding tendencies (disseminated intravascular coagulation (DIC), internal hemorrhage, etc.).
11. Ascites or pleural fluid requiring active medical management including paracentesis, or hyponatremia (defined as serum sodium value of < 130 mEq/L).
12. Patients who have been administered a drug in a clinical trial or an unapproved drug within three months before enrollment.
13. Patients who have previously treated with the test drug (rigosertib sodium).
14. Patients with known allergy to polyethylene glycol or gelatin capsules.
15. Patients with an addiction to a legal or illegal drug, or with alcohol dependency.
16. Patients who are pregnant or may become pregnant, or lactating mothers.
17. Patients who have not consented to the following contraceptive measures. Patients will avoid sexual intercourse with sexual partners or should use the following contraceptive methods in these time periods: for male patients during the administration period of the trial and for six months after the end of administration; female patients during the administration period of the trial, and until a second menstrual period is confirmed after the end of administration (or in the case of female patients with no menstrual period, for two months after the end of administration).

    * Male patients: Patients will always use a condom. For effective contraception, it is recommended that the female partner also use the contraceptive methods for female patients.
    * Female patients: Female patients who may become pregnant should use one or more types of the following contraceptive methods. In addition, the male partner will always use a condom. Oral contraceptive (birth control pills) , Intrauterine device (IUD) , Tubal ligation
18. Other patients judged to be unsuitable by an investigator or sub-investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Goto, Study Director — SymBio Pharmaceuticals
Locations (4):
- Japan (4):
  - Research site, Nagoya, Aichi-ken
  - Research site, Isehara, Kanagawa
  - Research site, Sendai, Miyagi
  - Research site, Kyoto

RESULTS

PARTICIPANT FLOW:
Groups:
- SyB C-1101 280 mg/Dose Group: Cohort 1: Participants were administered 280 mg/dose of SyB C-1101 twice daily orally for 14 consecutive days, followed by 7-day observation period.
  The treatment period of 21 days constitutes 1 cycle, and the treatment was allowed for up to cycles.
  The participants received SyB C-1101 only once daily on Day 1 and Day 14 of Cycle 1 for the investigation of the pharmacokinetics.
- SyB C-1101 560 mg/Dose Group: Cohort 2: Participants were administered 560 mg/dose of SyB C-1101 twice daily orally for 14 consecutive days, followed by 7-day observation period.
  The treatment period of 21 days constitutes 1 cycle, and the treatment was allowed for up to cycles.
  The participants received SyB C-1101 only once daily on Day 1 and Day 14 of Cycle 1 for the investigation of the pharmacokinetics.
Period: Overall Study
Arm/Group | SyB C-1101 280 mg/Dose Group | SyB C-1101 560 mg/Dose Group
Started | 3 | 6
Completed | 2 | 5
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who received at least 1 dose of SyB C-1101 either at 280 mg/dose or 560 mg/dose orally.
Arm/Group | All Participants
Number analyzed (Participants) | 9
Age, Customized [Number; unit: participants]
  50-59 years | 1
  60-69 years | 3
  70-79 years | 4
  80- years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Total Number Affected by Any Adverse Event (Details are presented in Adverse Event section)
Time Frame: Up to 18 weeks
Measure: Number; unit: participants
Arm/Group | SyB C-1101 280 mg/Dose Group | SyB C-1101 560 mg/Dose Group
Number analyzed (Participants) | 3 | 6
participants | 3 | 6

2. Primary Outcome: Number of Participants Who Experienced Dose-limiting Toxicities (DLTs)
Description: A DLT was defined as adverse events for which a causal relationship with the investigational drug could not be ruled out and which met the following criteria that occurred by the final observation in Cycle 1. DLTs were also assessed in the Efficacy and Safety Assessment Committee.
  Criteria
  1. Grade 3 or higher non-hematologic toxicity. However, nausea, vomiting, diarrhoea, pyrexia, stomatitis, and esophagitis/dysphagia are excluded (Grade 3 nausea, vomiting, diarrhoea, and pyrexia that cannot be controlled with antiemetic, antidiarrheal, or antifebrile agents are regarded as DLTs)
  2. Grade 3 or higher stomatitis, esophagitis, and dysphagia that persist for >= 4 days
Time Frame: Up to 21 days
Measure: Number; unit: participants
Arm/Group | SyB C-1101 280 mg/Dose Group | SyB C-1101 560 mg/Dose Group
Number analyzed (Participants) | 3 | 6
participants | 1 | 2

3. Secondary Outcome: Hematologic Remission Effect (IWG 2006 Criteria, Responses Sustained >= 4 Weeks)
Description: Definition
  Complete remission (CR) Bone marrow: <= 5% myeloblasts; normal maturation of all cell lines Peripheral blood: Hemoglobin (Hgb) >= 11 g/dL, Platelets >= 100×10^9/L, Neutrophils >= 1.0×10^9/L, Blasts 0%
  Partial remission (PR) Same as CR except bone marrow blasts decreased by >= 50% over pretreatment but still > 5%
  Marrow CR Bone marrow: <= 5% myeloblasts and decrease by >= 50% over pretreatment Peripheral blood: will be noted in addition to marrow CR
  Stable disease Failure to achieve at least PR, but no evidence of progression for > 8 weeks Disease progression
  Patients with:
  Less than 5% blasts: >= 50% increase in blasts to > 5% blasts 5%-10% blasts: >= 50% increase to > 10% blasts 10%-20% blasts: >= 50% increase to > 20% blasts 20%-30% blasts: >= 50% increase to > 30% blasts
  Any of the following:
  At least 50% decrement from maximum remission/response in granulocytes or platelets Reduction in Hgb by >= 2 g/dL Transfusion dependence
Time Frame: Up to 60 weeks
Measure: Number; unit: participants
Arm/Group | SyB C-1101 280 mg/Dose Group | SyB C-1101 560 mg/Dose Group
Number analyzed (Participants) | 3 | 6
participants
  CR | 0 | 0
  PR | 0 | 0
  Marrow CR | 1 | 0
  Stable disease (SD) | 1 | 1
  Treatment failure | 0 | 0
  Disease progression | 0 | 3
  Not assessable | 1 | 2
  Remission rate | 1 | 0

4. Secondary Outcome: Hematologic Improvement Effect (IWG 2006 Criteria, Responses Must Last at Least 8 Weeks)
Description: Definition
  Hematologic Improvement Erythrocyte (HI-E):
  Hgb increase by >= 1.5 g/dL Relevant reduction of units of red blood cell (RBC) transfusions by an absolute number of at least 4 RBC transfusions/8 week compared with the pretreatment transfusion number in the previous 8 week. Only RBC transfusions given for a Hgb of <= 9.0 g/dL pretreatment will count in the RBC transfusion response evaluation
  Hematologic Improvement Platelet (HI-P):
  Absolute increase of >= 30×10^9/L for patients starting with > 20×10^9/L platelets Increase from < 20×10^9/L to > 20×10^9/L and by at least 100%
  Hematologic Improvement Neutrophil (HI-N):
  At least 100% increase and an absolute increase > 0.5×10^9/L
  Progressive disease / Relapse:
  At least 1 of the following:
  At least 50% decrement from maximum response levels in granulocytes or platelets Reduction in Hgb by >= 1.5 g/dL Transfusion dependence
Time Frame: Up to 18 weeks
Measure: Number; unit: participants
Arm/Group | SyB C-1101 280 mg/Dose Group | SyB C-1101 560 mg/Dose Group
Number analyzed (Participants) | 3 | 6
participants
  HI-E | 0 | 0
  HI-P | 1 | 0
  HI-N | 0 | 0
  Progressive disease | 0 | 1
  Relapse | 0 | 0
  Not assessable | 2 | 5
  Hematologic improvement rate | 1 | 0

5. Other Pre Specified Outcome: Maximum Tolerated Dose (MTD)
Description: MTD was investigated with an index of DLT
Time Frame: Up to 18 weeks
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 9
participants | NA — MTD was not reached

ADVERSE EVENTS:
Time Frame: Up to 18 weeks for each dosing cohort
Description: All participants who received at least one dose of SyB C-1101.
Arm/Group | SyB C-1101 280 mg/Dose Group | SyB C-1101 560 mg/Dose Group
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SyB C-1101 280 mg/Dose Group (N=3) | SyB C-1101 560 mg/Dose Group (N=6)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SyB C-1101 280 mg/Dose Group (N=3) | SyB C-1101 560 mg/Dose Group (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (2) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Reticulocyte count decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No